CLINICAL TRIAL: NCT06207994
Title: Evaluation of the Impact of a Narrower SpO2 Target Range on Performance of an Automatic FiO2 Control System: a Randomized Study
Brief Title: PRICO: OPTI Target Range
Acronym: POSTR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Czech Technical University in Prague (Other)
Collaborators: University Hospital, Motol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PricoOptiTR
Record Dates: First submitted 2023-12-18; First posted 2024-01-17 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Neonatal Respiratory Distress; Very Low Birth Weight Infant
Keywords: SpO2 Target Range; pulse oximetry; automatic oxygen control
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: Subjects will be switched between the standard target range, the narrow target range, and the target range with a higher median every 12 hours. The sequence will be randomized differently for each subject, with a balanced block design such that every 3 days each range is evaluated twice.
  Once enrolled, each subject will continue in the study with regular changes in averaging time through the course of their need for A-FiO2 or 30 days, whichever is shorter. All other elements of care will be as routinely used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Target Range (No Intervention): The SpO2 TR width is set to 5% SpO2, as is routine in the department. The actual TR will vary depending on the GA, as is standard practice in the department.
- Narrow Target Range (Experimental): The SpO2 TR width is set narrower than the Standard TR. The actual TR will vary depending on the GA, as is standard practice in the department.
  Interventions: Device: Narrow TR
- Shifted Target Range (Experimental): The SpO2 TR width is set as the Standard TR. The median of the TR is shifted up compared to the Standard TR. The actual TR will vary depending on the GA, as is standard practice in the department.
  Interventions: Device: Shifted TR

INTERVENTIONS:
Device: Narrow TR — The width of the PRICO SpO2 TR is set to 3% SpO2.
  Arms: Narrow Target Range
Device: Shifted TR — The lower and the upper limits of the PRICO SpO2 TR are increased by 1% SpO2.
  Arms: Shifted Target Range

SUMMARY:
The aim of the study is to determine if a narrower SpO2 Target Range setting automated control of FiO2 (A-FiO2) is more effective than a wider SpO2 Target Range

DETAILED DESCRIPTION:
A-FiO2 systems have consistently proven to be more effective than manual control. Because it is more precise than manual control, studies of some A-FiO2 systems found small differences in the set target range (shift in the median and width) can optimize the relative performance. Similar studies of the A-FiO2 system (PRICO) used in the investigator's NICU have not been conducted.

The standard of practice in the investigator's NICU is to use 4 different target ranges to balance the risk of hypoxia and hyperoxia based on the gestational age vulnerabilities. Based on the studies of other A-FiO2 systems the investigators believe a slightly narrower width target range would be more effective. Therefore, a small systematic study is needed to determine the optimal set target range to achieve the therapeutic goal.

ELIGIBILITY:
Inclusion Criteria:

* All VLBW on respiratory support and oxygen requirements after 2 weeks of age in the NICU are eligible after informed consent is obtained.

Exclusion Criteria:

* Informed consent is not obtained
* Recording device for automated control of FiO2 is not available

Min Age: 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Percent time in the set SpO2 target range | 30 days of intervention if possible
  Percent time in the set SpO2 target range (compliance). Periods with SpO2 higher than the target range with FiO2 = 0.21 will be included in the target range compliance.
Percent time at SpO2 ≤80% and >98% | 30 days of intervention if possible
  Percent time at SpO2 ≤80% and >98% (safety). Periods with SpO2 higher than 98% with FiO2 = 0.21 will be excluded.

SECONDARY OUTCOMES:
Percent time above the set SpO2 target range | 30 days of intervention if possible
  Percent time above the set SpO2 target range. Periods with SpO2 higher than the target range with FiO2 = 0.21 will be excluded from time above the target range.
Percent time below the set SpO2 target range | 30 days of intervention if possible
  Percent time below the set SpO2 target range.

OTHER OUTCOMES:
Associated effects | 30 days of intervention if possible
  Effects associated with the mode of ventilation and set SpO2 control (based on gestational age) will be explored. The effects will be treated as covariables in a multivariate linear regression model with SpO2 target range compliance as a dependent variable.
Stability | 30 days of intervention if possible
  Effects associated with infant stability will be explored. The stability will be assessed based on the mean time in the SpO2 target range.

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Orlova, MD, Principal Investigator — Motol University Hospital Prague, Neonatal Unit; Jan Janota, MD, PhD, Principal Investigator — Motol University Hospital Prague, Neonatal Unit; Thomas E Bachman, MSc, Principal Investigator — Czech Technical University in Prague; Jana Dornakova, MD, Principal Investigator — Motol University Hospital Prague, Neonatal Unit
Locations (1):
- Motol University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be made available upon reasonable request in a deidentified, HIPAA-compliant form.